CLINICAL TRIAL: NCT05602376
Title: Improving HIV Testing, Linkage, and Retention in Care for Men Through U=U Messaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Desmond Tutu HIV Foundation (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Institutes of Health (NIH) (NIH); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R01MH129223 (NIH); R01MH129223 (NIH)
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: HIV Infections; Men; Treatment Adherence
Keywords: HIV; HIV testing; Men; U=U; Viral suppression; Treatment as Prevention; Viral load; ART uptake; Undetectable; Untransmittable
MeSH Terms: conditions — HIV Infections; Multiple Endocrine Neoplasia Type 1; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Two hybrid type 1 effectiveness-implementation randomized controlled trials to evaluate the impact of U=U messages on men's uptake of community-based HIV testing and treatment initiation (Aim 1), and achievement of viral suppression (Aim 2)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Aim 1: Site-testing-days will be randomised 1:1 to implement either U=U (intervention) or SoC (Control) messaging scripts for both invitation-to-test and ART initiation.
  Aim 2: Randomization will be stratified by the 6 study clinics, to account for possible differences in the baseline viral loads of the catchment area populations initiating ART within each clinic with individual-level randomization will be used with random block sizes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- U=U testing messaging scripts (Experimental): Aim 1: Human-centred designed, behavioural nudge theory informed U=U messaging intervention to improve HIV testing uptake by men
  Interventions: Behavioral: U=U testing messaging scripts
- U=U adherence messaging scripts (Experimental): Aim 2: Human-centred designed, behavioural nudge theory informed U=U messaging intervention to improve ART adherence, HIV viral suppression and retention in care
  Interventions: Behavioral: U=U adherence messaging scripts
- Standard of Care (SoC) messaging (No Intervention): Aim 1: SoC messaging scripts will be used to both invite men for CB-HTS and to refer those that test HIV-positive for DoH clinic-based ART initiation
  Aim 2: SoC messaging as part of ART initiation counselling, and as part of their HIV care and treatment program

INTERVENTIONS:
Behavioral: U=U testing messaging scripts — On site testing days randomized to the intervention, trained health promoters employed by the mobile testing venues will use U=U messaging scripts to invite men in the vicinity to seek HIV testing services on that day. On intervention days, the U=U messaging will also be used by counselors at the testing venue when referring those who test HIV positive to clinic-based ART initiation services provided by the local Department of Health
  Arms: U=U testing messaging scripts
Behavioral: U=U adherence messaging scripts — After receiving standard ART initiation and adherence counselling from a DoH clinic nurse per South African National Guidelines, RCs will deliver a U=U message and hand participants a small business card with a brief U=U message on it. Participants will then receive monthly SMS booster messages (but can opt out) and monthly in-clinic booster messages during routine medical refill visits, again with a business card for messaging reinforcement.
  Arms: U=U adherence messaging scripts

SUMMARY:
This study will evaluate the impact of U=U messaging and counseling on gaps in the HIV care cascade for men, including testing uptake and ART initiation (Aim 1), achieving viral suppression and retention in care (Aim 2) in two provinces in South Africa. The U=U message communicates the compelling idea that PLHIV who take ART and have an undetectable viral load (<200 copies/mL) cannot sexually transmit HIV. Additionally, the investigators will conduct a multi-method evaluation to inform future implementation of U=U messaging interventions (Aim 3).

DETAILED DESCRIPTION:
Increasing the coverage of HIV testing and treatment among people living with HIV (PLHIV) is essential for ending the global AIDS epidemic. Unfortunately, compared to women, men living with HIV (MLHIV) are less likely to know their HIV status, start anti retroviral treatment, or achieve viral suppression. Given that new HIV infections among women are driven, in part, by men's testing and treatment gaps, reducing the gender gap in testing uptake, treatment initiation and achievement of viral suppression by men must be prioritized in order to accelerate the decline in HIV incidence among women, improve men's HIV-related health outcomes and achieve the UNAIDS 95-95-95 goals by 2030.

In this study, the investigators evaluate the effectiveness of Undetectable Equals Untransmittable or "U=U" messaging for closing the gender gap in the HIV cascade. Particularly for men, the U=U message has the potential to accelerate progress towards the 95-95-95 targets by: 1) reducing anxiety associated with HIV testing (1st 95); 2) encouraging people who test HIV positive to initiate ART (2nd 95); and 3) reducing fear of transmitting HIV to sexual partners by promoting treatment adherence to achieve viral suppression (3rd 95). While there is a growing knowledge of Treatment as Prevention (TasP)/U=U among PLWH in Western countries, the reach and penetration of the U=U message in sub-Saharan Africa has been limited and few studies have tested the impacted of accessible U=U messages on ART uptake and adherence in sub-Saharan Africa.

Building on the investigators prior work on U=U messaging informed by behavioral economics and human-centered design, they propose to conduct two hybrid type 1 effectiveness-implementation randomized controlled trials to evaluate the impact of U=U messages on men's uptake of community-based HIV testing and treatment initiation (Aim 1), and achievement of viral suppression (Aim 2). The investigators will also conduct a multi-method evaluation to inform future implementation of U=U messaging interventions. To improve the generalizability of the findings, the study will be conducted in two provinces in South Africa (Western and Eastern Cape). If effective, the intervention can shape global HIV testing and treatment counselling guidelines and practices. The expert, multi-institutional collaborations will allow for the application of previous research findings, leverage unique implementation platforms and resources, and rapidly disseminate the findings.

ELIGIBILITY:
Inclusion Criteria:

AIM 1:

1. male
2. aged ≥15 years
3. present a study issued invitation card to site receptionist
4. ability to provide informed consent.

AIM 2:

1. cis-gender men
2. aged ≥15 years
3. newly initiating ART (i.e., treatment naïve) or re-initiating ART after 6 months of being lost-to-care
4. live in Buffalo City or Cape Town Metro Health Districts
5. provide written informed consent

Min Age: 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3642 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
ART initiation among those invited to test for HIV | 30-day follow-up period
  Proportions of ART initiation among all people invited to test in each study arm over the year of Aim 1 data collection
Proportion with viral load suppression | 6-month visit
  Proportions of people who have documented viral suppression at the 6-month visit in each study arm during Aim 2

SECONDARY OUTCOMES:
% who agree to testing | Baseline
  Proportions of testing uptake among all people invited to test in each study arm over the year of Aim 1 enrolment.
Proportion retained in care | 12-month visit
  Proportions of people who have a recorded viral load at their 12-month visit in each study arm during Aim 2.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Medina-Marino, PhD, Principal Investigator — Desmond Tutu Health Foundation; Alison Buttenheim, PhD, MBA, Principal Investigator — Penn Nursing and Perelman School of Medicine, University of Pennsylvania
Locations (2):
- South Africa (2):
  - Buffalo City Metro, East London, Eastern Cape
  - Cape Town Metro, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, Analytic Code
Access Criteria: Based on contractual agreement

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-10-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT05602376/SAP_000.pdf